CLINICAL TRIAL: NCT06786923
Title: The Effect of Transcutaneous Auricular Vagus Nerve Stimulation on the Incidence of Delayed Gastric Emptying After Pancreatoduodenectomy: A Randomized Controlled Trial
Brief Title: The Effect of taVNS on the Prognosis of Patients Undergoing Pancreatoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Chaochao Zhong, Principal Investigator, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-K265-02
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Delayed Gastric Emptying
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous auricular vagus nerve stimulation (taVNS group) (Experimental): Patients in the taVNS group will have a transcutaneous auricular vagus nerve stimulation device with a transparent, non-insulated thin film placed on the cymba conchae of the left ear. TaVNS will be administered on the day of surgery (starting 30 minutes before anesthesia induction and continuing until the end of the surgery, terminating after the removal of the endotracheal tube in the PACU). The stimulation parameters are set as follows: frequency 25 Hz, pulse width 200 μs, 30 seconds on / 30 seconds off, with the current intensity set to the maximum amplitude the patient can tolerate (just below the pain threshold).
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulator
- Sham transcutaneous auricular vagus nerve stimulation (Sham taVNS group) (No Intervention): Patients in the Sham taVNS group will have a transcutaneous auricular vagus nerve stimulation device with a transparent insulating film placed on the cymba conchae of the left ear on the day of surgery. The stimulation parameters, method, and duration will be the same as those in the taVNS group. However, due to the insulating film applied to the stimulation device in the sham group, patients will not actually receive any stimulation.

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulator — Intervention Timing of Transcutaneous Auricular Vagus Nerve Stimulator: The intervention will begin 30 minutes before anesthesia induction and continue until the end of the surgery, terminating after the removal of the endotracheal tube in the PACU. The stimulation parameters are set as follows: frequency 25 Hz, pulse width 200 μs, 30 seconds on / 30 seconds off, with the current intensity set to the maximum amplitude the patient can tolerate (just below the pain threshold).
  Arms: Transcutaneous auricular vagus nerve stimulation (taVNS group)

SUMMARY:
To explore the effects of transcutaneous auricular vagus nerve stimulation (taVNS) during the perioperative period on the incidence of delayed gastric emptying after pancreatoduodenectomy and its possible mechanisms.

DETAILED DESCRIPTION:
Patients are recruited one week prior to the start of the trial, during which they are informed about the experimental protocol and associated risks. After obtaining informed consent and signatures, they are enrolled as study participants. Patients who meet the trial criteria are randomly assigned in a 1:1 ratio to the control group (sham taVNS group) and the intervention group (taVNS group, with taVNS intervention starting 30 minutes prior to anesthesia induction and continuing until the end of surgery, terminating after the removal of the endotracheal tube in the PACU), in a double-blind manner (with taVNS intervention and postoperative follow-up conducted by different researchers).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosed with pancreatic tumors or periampullary tumors by imaging or pathology and scheduled for pancreaticoduodenectomy;
* No distant metastases and tumors are resectable;
* Classified as American Society of Anesthesiologists (ASA) physical status I to III;
* Capable of understanding the study procedures and various assessment scales and able to effectively communicate with the researchers;
* Willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* Patients with other malignant tumors;
* Patients who have undergone chemotherapy or radiotherapy before surgery;
* Patients with chronic organ dysfunction;
* Patients with a history of gastrectomy or other gastric surgeries;
* Patients diagnosed with chronic gastrointestinal inflammation, peptic ulcers, or a history of gastroparesis, pyloric, or other gastrointestinal obstructions;
* Patients with a history of autonomic dysfunction (e.g., peripheral neuropathy, vagotomy, thyroid dysfunction, amyloidosis, asthma, heart failure, renal dysfunction, or alcoholism);
* Patients with implanted stimulators (e.g., pacemakers, implanted vagus nerve stimulators, deep brain stimulators, spinal cord stimulators), cochlear implants, or metallic implants (excluding dental work);
* Patients who recently used prokinetic agents, cholinergic or anticholinergic drugs, or hormones;
* Patients who received vagus nerve stimulation or acupuncture within 1 month before the study;
* Patients with skin damage or dermatological conditions at the stimulation site;
* Patients with a preoperative heart rate below 60 beats per minute;
* Patients unable to cooperate with assessments;
* Patients participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Delayed Gastric Emptying | The first 7 days postoperatively
  The definition of delayed gastric emptying (DGE) after pancreatic surgery, as suggested by the International Study Group of Pancreatic Surgery (ISGPS), is as follows:
  Excluding mechanical factors such as intestinal obstruction and anastomotic stricture, DGE can be diagnosed if any of the following conditions are met:
  1. The need for nasogastric tube placement persists for more than 3 days postoperatively.
  2. Re-insertion of the nasogastric tube is required due to vomiting or other reasons after its removal.
  3. The patient is unable to consume solid food 7 days postoperatively.

SECONDARY OUTCOMES:
Incidence of Grade A, B, and C Postoperative Delayed Gastric Emptying | The first 21 days postoperatively
  Based on the severity of postoperative delayed gastric emptying (DGE) following pancreatic surgery, DGE is classified into three grades: A, B, and C:
  Grade A: Requires nasogastric tube placement from postoperative days 4 to 7 or re-insertion of the tube after 3 days. Patients are unable to tolerate oral solid food for more than 7 days postoperatively.
  Grade B: Requires nasogastric tube placement from postoperative days 8 to 14 or re-insertion of the tube after 7 days. Patients are unable to tolerate oral solid food for more than 14 days postoperatively.
  Grade C: Nasogastric tube cannot be removed within 14 days postoperatively or requires re-insertion after 14 days. Patients are unable to tolerate oral solid food for more than 21 days postoperatively.
Duration of Nasogastric Tube Drainage After Surgery | Up to 3 weeks postoperatively
  The time from the end of surgery to the first removal of the nasogastric tube
Time to First Intake of Solid Food | Up to 3 weeks postoperatively
  The time to the first intake of solid food after surgery
Incidence of Other Postoperative Complications Following Pancreatic Surgery (Including Pancreatic Fistula, Bile Leakage, Chylous Fistula, Postoperative Bleeding, and Abdominal Infection) | Up to 5 weeks postoperatively
  Incidence of other postoperative complications after pancreatic surgery (such as pancreatic fistula, bile leak, chyle leak, postoperative bleeding, and intra-abdominal infection)
Severity of Postoperative Complications (Assessed Using the Clavien-Dindo Classification System) | Up to 5 weeks postoperatively
  The severity of postoperative complications (assessed using the Clavien-Dindo classification) refers to a system that classifies postoperative complications based on their severity. The Clavien-Dindo classification system is a widely used standardized method in clinical practice, designed to help doctors objectively assess the severity of postoperative complications, providing a basis for clinical management and research.The system classifies postoperative complications into five levels based on severity, ranging from Grade I (mildest) to Grade V (most severe). Each grade represents the impact of the complication on the patient and the degree of treatment required.
Total Length of Hospital Stay | Up to 5 weeks postoperatively
  The total length of hospital stay refers to the entire duration of the patient's hospitalization from admission to discharge.
NRS Score Measured on the Day Before Surgery, and Postoperative Days 1, 3, and 7 | Preoperative Day 1, Postoperative Day 1, 3, 7
  The NRS (Numerical Rating Scale) is used to assess the intensity of pain.The higher the score, the more severe the pain.
Hospital Anxiety and Depression Scale (HADS) Before Surgery and on Postoperative Days 7 and 14 | Preoperative Day 1, Postoperative Day 7, 14
  The Hospital Anxiety and Depression Scale (HADS) is used to evaluate the severity of anxiety and depression in individuals.
PROMIS SD-SF 8a Assessment on Preoperative and Postoperative Days 7 and 14 | Preoperative Day 1, Postoperative Day 7, 14
  The Patient-Reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8a (PROMIS SD-SF 8a) is an 8-item self-reported questionnaire developed by the Patient-Reported Outcomes Measurement Information System to assess sleep disturbance over the past 7 days. It evaluates aspects such as difficulty falling asleep, sleep maintenance, sleep quality, and daytime functioning, providing a standardized measure of sleep disturbance severity.
Incidence of Postoperative Nausea and Vomiting (PONV) within 48 Hours | The first 48 hours postoperatively
  To determine the incidence of postoperative nausea and vomiting (PONV) within 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chao Zhong, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No